CLINICAL TRIAL: NCT03589521
Title: Adapting Alcohol Behavioral Couple Therapy for Service Members in Post-Deployment
Acronym: ABCT_Mil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Epstein, Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA023027; 5R34AA023027 (NIH)
Record Dates: First submitted 2018-06-08; First posted 2018-07-18 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Abuse
Keywords: Veterans; Cognitive Therapy; Couple Therapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABCT_Military (Experimental): ABCT_Military manual will address alcohol use, couple issues and military specific issues. Required interventions include: routine interventions, overview of treatment, reintegration issues, motivational techniques, patient-focused interventions for abstinence, partner-related interventions for abstinence, couple interventions, general coping skills, social skills and relapse prevention. In addition, to personalize each treatment plan, interventions from optional modules (e.g., intimate partner violence (IPV), depression, trauma, and traumatic brain injury (TBI)) will be integrated into each couple's treatment plan depending on clinical presentation.
  Interventions: Behavioral: ABCT_Military

INTERVENTIONS:
Behavioral: ABCT_Military — 15 Weekly Couple Therapy Sessions

SUMMARY:
The specific aims of the ABCT_Military project are as follows: 1) To modify the existing, Alcohol Behavioral Couple Therapy (ABCT) model to treat service members in the reconstitution (post deployment, reintegration, or separation) stage of service, and develop optional psychoeducation modules to address relevant co-morbid problems and challenges in this population in a weekly, 15 session, stand-alone outpatient format. 2) To test feasibility and preliminary efficacy of the study intervention protocol in a successive cohort design for one cohort of 8 couples and one cohort of 22 couples, with iterative manual revision.

DETAILED DESCRIPTION:
The study staff will screen potential participants over the phone, and arrange Baseline (BL) research interviews for appropriate couples. The couple will meet with the program interviewer for approximately 2 hours. After the BL interview, couples will be scheduled to attend therapy sessions. Couples will complete brief within treatment self-report assessments. Couples will complete a post treatment follow up interview four months after session 1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older;
* Married (or separated with efforts to reconcile) or in a committed relationship (cohabiting, or in an exclusive dating relationship), or significant other (SO) (first, second or third degree relative (including step relative or in-law) or close trusted friend not active in same military branch. The service member only must meet the following inclusion criteria:
* Served or serving in the U.S. Military,
* Current Alcohol Use Disorder diagnosis, or drink at high risk levels as defined by NIAAA (2010)

Exclusion Criteria:

* Either individual is not fluent in the English language.

Exclusion criteria for the service member only:

* Unstabilized Psychotic disorder in past six months

Exclusion criteria for both members of the couple if SO is spouse/romantic partner:

* Either partner is fearful of participating in couple therapy OR either partner suffered severe physical abuse from partner when perpetrator not intoxicated, in past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Percent Drinking Days (PDD) | Change from baseline at 4 months post Session 1
  Derived from Timeline Followback (TLFB)
Percent Heavy Drinking Days | Change from baseline at 4 months post Session 1
  Derived from Timeline Followback (TLFB)
Mean Drinks Per Drinking Day | Change from baseline at 4 months post Session 1
  Derived from Timeline Followback (TLFB)
Couple Satisfaction Inventory 16 | Change from baseline at 4 months post Session 1
  16 item measure assessing satisfaction in couple relationship. Scores range from 0 to 81 and higher scores indicate higher levels of relationship satisfaction. Total score is calculated by summing all values.

SECONDARY OUTCOMES:
Coping Strategies Scale | Change from baseline at 4 months post Session 1
  25-item brief measure assessing coping in alcohol-specific and non-alcohol situations. Scores range from 1-4 and higher scores indicate greater use of coping skills. Total score is calculated by averaging all values.
World Health Quality of Life Questionnaire - Bref | Change from baseline at 4 months post Session 1
  26-item self report assessing quality of life across 4 domains/subscales: Physical health, Psychological, Social relationships, Environment. The first two items measure quality of life and overall health and are examined separately, with scores ranging from 1-5. The four domain scores are calculated by averaging values and scores range from 1-5. Higher scores indicate higher quality of life within each domain. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100 (full scale measure).
Treatment Services Review | Weekly during treatment, for up to 16 weeks
  Interview assessing quantity and type of services received (e.g., health, psychological) outside of study intervention. Total scores are calculated by summing the number of outside services used. Total scores have a minimum of 0 and no maximum value.
Working Alliance Inventory Short Form | Baseline and through study completion, about 16 weeks
  12-item self-report measure of the therapeutic alliance. Total scales are calculated by summing all values. Values range from 1-7 with total scores ranging from 12 to 84). Higher scores indicate greater alliance.
Post-Traumatic Stress Disorder (PTSD) | Baseline
  Percent of sample with a PTSD diagnosis as determined by scores on the Life Events Checklist (LEC-5) and the PTSD Checklist (PCL-5).
PTSD Checklist (PCL-5) | Baseline and through study completion, about 16 weeks
  20-item self-report questionnaires assessing current symptoms of PTSD, used to assess current (past 30 days) PTSD severity. Total scores are calculated by summing all values. Scores on the PCL-5 range from 0-80 and reflect a global PTSD severity score, with higher scores indicating greater severity.
Use of Treatment Skills | Baseline and through study completion, about 16 weeks
  Self-report questionnaire assessing use of skills learned during treatment. Item scores range from 1-5 and a total score is calculated by summing all values. Higher scores indicate greater use of skills.

OTHER OUTCOMES:
Beck Depression Inventory II (BDI-II) | Change from baseline at 4 months post Session 1
  self-report questionnaire assessing depression symptoms over the prior two weeks (scores range 0-63) and higher scores indicate greater depression symptomatology. All item scores are summed to attain a total score.
Copello Coping Questionnaire | Change from baseline at 4 months post Session 1
  30 item self-report assessing partner alcohol-related coping skill use. Total score is calculated by summing the values from each item and scores range from 0-90 with higher scored indicating greater use of coping strategies.
Intimate Partner Violence (IPV) | Change from baseline at 4 months post Session 1
  Percent of sample with IPV as determined by scores on the Conflict Screener Form H.
Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) Short Form | Change from baseline at 4 months post Session 1
  19 item self-report questionnaire assessing client readiness for change. An additional item assesses the client's motivation for coming to therapy. There are three sub scales (Recognition, Ambivalence, and Taking Steps) which are derived from individual items. Higher scores indicate greater recognition, ambivalence and taking steps and scores range from 7 to 35, 4 to 20, and 8-40, respectively.
Traumatic Brain Injury (TBI) | Baseline
  Percent of sample with a TBI as determined by scores on the TBI Checklist.
Traumatic Brain Injury (TBI) Checklist | Change from baseline at 4 months post Session 1
  Severity of TBI as determined by total scores on the TBI Checklist. Scores are calculated by summing individual item scores with possible scores ranging from 8 to 88.
Partner Quantity Frequency Questionnaire | Change from baseline at 4 months post Session 1
  Self-report questionnaire assessing frequency and quantity of current and lifetime substance use. Measure is used to provide descriptive data about partner substance use. Total scores are not used.
Medical History Questionnaire | Change from baseline at 4 months post Session 1
  40 item self-report assessing presence of medical conditions currently and in the past. Scores are calculated by summing individual item scores with possible scores ranging from 0 to 40. Higher scores indicate greater number of medical problems.
End of Treatment Questionnaire | 4 months post session 1
  Self-report questionnaire of helpfulness of therapy elements on a 7 point scale of -3 (greatly harmful), -2, -1, 0 (neutral), +1, +2, +3 (greatly helpful). Total scores are calculated by averaging scores across individual items.
Brief COPE | Change from baseline at 4 months post Session 1
  28 item self-report assessing general coping skill use. Sub scale scores are calculated by summing individual items (2 items per sub scale) with possible scores of 2 to 8. The sub scales are: Self-distraction, Active coping, Denial, Substance use, Use of emotional support, Use of instrumental support, Behavioral disengagement, Venting, Positive reframing, Planning, Humor, Acceptance, Religion, and Self-blame. Higher scores reflect greater use of each category of coping skills.
Client Satisfaction Questionnaire | 4 months post session 1
  8 item self-report assessing satisfaction with treatment. Individual item scores are averaged to calculate a total score with possible scores ranging from 0 to 4. Two additional items assessed the client's ideal number of sessions and length of treatment, with scores ranging from 1 to 24 sessions and 1-12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Epstein, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with investigators outside of the core study team.